CLINICAL TRIAL: NCT04079491
Title: Dental Hygienists and Oral Mucosal Inspection - Extent, Knowledge and Perceived Barriers
Brief Title: Intra and Extra Oral Inspection of Oral Mucosa
Status: Terminated | Type: Observational
Why Stopped: Poor responce
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Kristina Edman, Principal Investigator, Dalarna County Council, Sweden
Other Study IDs: Inspection oral mucosa
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Oral Lichen Planus; Oral Leukoplakia; Erythroplakia
Keywords: oral mucosal lesions; dental hygienist
MeSH Terms: conditions — Lichen Planus, Oral; Leukoplakia, Oral; Erythroplasia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dental hygienists: all dental hygienists members in the trade union for dental hygienists
  Interventions: Other: questionnaire survey

INTERVENTIONS:
Other: questionnaire survey — A web-based questionnaire will be send by the trade union for dental hygienists

SUMMARY:
Dental health professionals have a responsibility to perform routine intra- and extraoral inspection on their patients for detecting abnormalities. As dental hygienists (DH) and dentist (D) often see their patients on a regular basis, they have the opportunity to provide this screening, and at an early stage detect abnormalities.

DETAILED DESCRIPTION:
In Sweden, education and training in intraoral inspection of the oral mucosa is a part of the curriculum in dental hygienists education, so there is an expectation that the dental hygienist routinely perform tactile and visual intraoral inspections in practice. However, DH are not trained in extra oral inspection and are not allowed to diagnose an oral mucosal lesion, but are trained to identify abnormalities and determine whether the patient needs referral to a dentist. It is also to expect that the DH are capable to identify risk behaviors, such as alcohol and smoking, and recommend, and offer smoking cessation or refer the patient to a certified profession for smoking cessation.

In 2007, The World Health Assembly (WHA) adopted a resolution to prevent oral cancer. The resolution urged the member states to ensure that measures against oral cancer was integrated into a national cancer control program by engaging and train dental personnel in screening, early diagnosis and treatment. Oral cancer is a severe oral health issue as it is potentially fatal and is the 5-6 most common tumor with approximately 275,000 cases for oral and 130,300 cases for pharyngeal cancers, excluding nasopharynx, globally. In Sweden,1000 new cases yearly is discovered and it is increasing. The explanation is an aging population and an increase in tonsil and tongue cancers caused by HPV, especially in younger subjects. Tumors caused by tobacco and alcohol are constant [7-9]. Despite the decreasing prevalence of smoking and certain smoking-associated cancers, an increased incidence of tonsillar cancer has been seen in both Finland and Sweden. High risk HPV (hrHPV) oral cancer is also increasing. The 5 year survival of oral cancer in Sweden is 55 % and only 3-4% in advanced cases. The etiology is hrHPV, exposure to tobacco and alcohol in 65% [13] and poor dental status. All are lifestyle factors so there are many opportunities for prevention and intervention. In 2016, 352 individuals in Sweden died in oral cancer compared with 135 individuals who died of cervical cancer. Leukoplakia (LP), erythroplakia (EP) and oral lichen planus (OLP) are the dominating oral premalignant entities. The diagnosis are clinical and often by biopsies. The nonhomogeneous have a risk of malignant transformation of 3.6-8.9% in Scandinavia. OLP is a chronic inflammatory lesion where the atrophic and erosive types have a risk of cancer development of 0.5-2%.

The potential for prevention is high, as the risk factors are well known. The Clinical examination discloses any potentially malignant lesions. Being aware of the increasing number of head, neck, and oral tumors we need to highlight the importance of inspection of the oral mucosa.

ELIGIBILITY:
Inclusion criteria:

* Registered dental hygienists members in the Swedish trade union

Exclusion criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All dental hygienists members in the trade union will be offered to participate
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Performance of intra and extra oral inspection of the oral mucosa | baseline
  A 27-item survey instrument using Likert-type and open-ended questions, constructed by dental hygienists and used in Canada, College of dental hygienists Nova Scotia, Canada is used. Frequency and comprehensiveness of intra- and extra-oral inspection is investigated and participants can answer always, usually, sometimes, rarely or never.
Barriers that might prevent dental hygienists from performing intra and oral inspection of the oral mucosa. | baseline
  From a drop down meny participants get seven alternative barriers; • Someone else in my office performs the exam [if selected drop down menu options appear: dentist, dental assistant, do not know, other
  * Lack of knowledge and/or skills to perform the exam
  * Lack of time
  * Concern about patient compliance
  * Concern over remuneration for services
  * Not sure if it is within the dental hygiene scope of practice
  * Other

CONTACTS AND LOCATIONS:
Overall Officials: Karin Gunnars Hellgren, Study Chair — Public Dental Health Region of Dalarna
Locations (1):
- Public Dental Service, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided